CLINICAL TRIAL: NCT04492410
Title: COVID-19 Infection Screening in Cancer Patients (NEOSCREENCOVID)
Acronym: NEOSCREENCOVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Antoine Lacassagne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2020/23; 2020-A01098-31 (Other: ANSM ID RCB)
Record Dates: First submitted 2020-07-28; First posted 2020-07-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2021-06

CONDITIONS: Cancer
Keywords: Covid-19; Screening
MeSH Terms: conditions — Neoplasms; COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental): screening using a rapid serological test with a drop of blood from a finger prick.
  Interventions: Other: rapid serological test

INTERVENTIONS:
Other: rapid serological test — screening using a rapid serological test with a drop of blood from a finger prick

SUMMARY:
Since December 2019, outbreak of COVID-19 caused by a novel virus SARS-Cov-2 has spread rapidly around the world and became a pandemic issue. Cancer patients seem to be at higher risk of infection and evolution to severe forms related to immunosuppression, according to the first published data from Chinese experience. However, the role of confounding factors such as age and smoking habits cannot be independently assessed. Supplementary data from a large retrospective Italian cohort suggest that the proportion of cancer patients with severe form of COVID-19 could be lower than expected. In addition, the proportion of asymptomatic SARS-Cov-2 infected cancer patients is unknown. Based on academic and expert's recommendations, most of cancer units have already modified cancer treatment during the pandemic, in order to limit the number of outpatient visits / inpatient admissions and then reduce or avoid cross infection of COVID-19, although the negative impact on patient's outcome (cancer recurrence or mortality) has not been established. Thus, a large screening for SARS-Cov-2 infection in treated cancer patients could help to: - Define an accurate prevalence of COVID-19 immunization in this population - Aggregate data on the relationship between clinical characteristics in cancer patients and COVID-19 risk. - Provide information about asymptomatic COVID-19 cases. - Organize effectively cancer units to separate infected and non-infected patients.

The RT-PCR gold-standard test for COVID-19 on nasal and pharyngeal swabs has limitations, as the test is not universally available, turnaround times can be lengthy, and reported sensitivities vary. It does not provide information about immunization status. Serological assays may be important for understanding the epidemiology of emerging SARS-Cov-2, including the burden and role of asymptomatic infections. Thus, the development of new devices or techniques for accurate diagnosis of SARS-CoV-2 infections, of fast and safe use, that could be spread in the local hospitals and clinics, would be a major advance for identifying and treating patients. In addition, information about the immunization of fragile people, such as cancer patients, could help to plan a safe strategy for anti-cancer treatment schedule and for the end of quarantine.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18-years old;
2. Patient treated for histologically proven cancer;
3. Patient that require at least one visit for anti-cancer treatment in a one-day outpatient care units
4. Patients that have previously been tested positive with a RT-PCR test from nasal swab that have been authorized to come to the hospital (after recovery or a 14-days quarantine period, according to local guidelines) can be included. 5. Patient willing and able to provide written informed consent/assent for the trial;

6. Patient affiliated with a health insurance system.

Exclusion Criteria:

1. Patient not able to give free consent
2. Patient not able to understand the protocol;
3. Patient not able to undergo the COVID-19 test
4. Vulnerable persons as defined by article L1121-5 - 8:

   1. Pregnant women, women in labour or breast-feeding mothers, persons deprived of their freedom by judicial or administrative decision, persons hospitalized without their consent by virtue of articles L. 3212-1 and L. 3213-1 and who are not subject to the provisions of article L. 1121-8
   2. Persons admitted to a social or health facility for reasons other than research
5. Adults subject to a legal protection order or unable to give their consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2020-07-21 (Actual); Primary Completion 2021-05-12 (Actual); Study Completion 2021-11-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the prevalence of COVID-19 | Day 1
  The rate of prevalence will be defined as the ratio of the number of positive patients to the number of patients tested based on the rapid serological test (presence of IgM and/or IgG).

SECONDARY OUTCOMES:
To evaluate patient's and health care professional's perception about the rapid serological test. | Day 1
  The assessment of the perception of the rapid serological test for patient and health care professional will be measured in terms of Pain, simplicity, rapidity and satisfaction, reported on a questionnaire:
  * • Pain: The pain assessment will be performed using a visual analog scale (VAS). The score will be graded between 0 (absence of pain) to 10 (maximum pain)
  * • Simplicity: The assessment of the satisfaction of care will be carried out using a Likert scale with 4 modalities. The score will be graded between "Poor" to "Very Good".
  * • Rapidity: The assessment of the satisfaction of care will be carried out using a Likert scale with 4 modalities. The score will be graded between "Poor" to "Very Good".
  * • Satisfaction with care: The assessment of the satisfaction of care will be carried out using a Likert scale with 4 modalities. The score will be graded between "Poor" to "Very Good"
To evaluate the concordance of COVID-19 positivity by the rapid serological test compared to the gold-standard RT-PCR on nasal swab for eligible patients | Day 1
  Diagnostic performance: sensibility, specificity, positive and negative predictive values, positive and negative likelihood ratio and area under the ROC curve, will be assessed to evaluate the rate of COVID-19 positive and COVID-19 negative serological rapid test on whole blood compared to the gold-standard RT-PCR on nasal swab.
To evaluate the concordance of COVID-19 positivity by the rapid serological test compared to a classic serological test (ELISA method) from whole blood | Day 1
  Diagnostic performance: sensibility, specificity, positive and negative predictive values, positive and negative likelihood ratio and area under the ROC curve, will be assessed to evaluate the rate of COVID-19 positive and COVID-19 negative serological rapid test on whole blood compared to an ELISA serological test on whole blood.
To evaluate the proportion of the patients who will have at least one positive testing among all the methods applied. | 6 months
  The rate of patients with at least one positive test among all the methods applied (rapid serological test and/or serological ELISA test and/or RT-PCR and/or ddPCR) will be defined.
To evaluate the number of patients who will get at least one new testing after the rapid serological test has been performed. | 6 months
  The proceedings of additional COVID-19 testing for corresponding patients will be described in terms of:
  * Time interval between the tests
  * Type and results of the subsequent tests
To compare the clinical and biological characteristics between positive and negative tested COVID-19 patients | 6 months
  The clinical and biological characteristics between positive and negative COVID-19 will be compared in term of:
  * Age, gender, BMI, performance status, smoking history, alcohol consumption, medical history and concomitant medication
  * clinical stage, location, type of treatment.
  * blood group, hematology, coagulation parameters and serum clinical chemistry
To describe the outcome of COVID-19 positive patients | 6 months
  The rate of hospital admission for severe COVID-19 form and death will be assessed.
To evaluate the impact of COVID-19 rapid serological test on the anti-cancer treatment schedule | 6 months
  A change on the anti-cancer treatment Schedule induced by the result of COVID-19 test will be defined as :
  * a medical treatment delay decision
  * or a treatment discontinuation decision

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Antoine Lacassagne, Nice, France

IPD SHARING:
Plan to Share IPD: No